CLINICAL TRIAL: NCT04657848
Title: Preliminary Efficacy Analysis of Cheng's Giraffe Reconstruction After Proximal Gastrectomy in Early Adenocarcinoma of Esophagogastric Junction : A Prospective Open-label Study
Brief Title: Preliminary Efficacy Analysis of Cheng's Giraffe Reconstruction After Proximal Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020361093
Record Dates: First submitted 2020-11-24; First posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Gastric Cancer; Reflux Esophagitis
Keywords: proximal gastrectomy, Cheng's Giraffe reconstruction
MeSH Terms: conditions — Stomach Neoplasms; Esophagitis, Peptic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- proximal gastrectomy combined with Cheng's Giraffe reconstruction (Experimental): proximal gastrectomy combined with gastric tube interposition esophagogastrostomy with reconstruction of His angle and fundus (Cheng's Giraffe reconstruction)
  Interventions: Procedure: proximal gastrectomy combined with Cheng's Giraffe reconstruction

INTERVENTIONS:
Procedure: proximal gastrectomy combined with Cheng's Giraffe reconstruction — proximal gastrectomy combined with gastric tube interposition esophagogastrostomy with reconstruction of His angle and fundus (Cheng's Giraffe reconstruction)

SUMMARY:
In the past years, the adenocarcinoma of the esophagogastric junction (AEG) has been increasing obviously in China. It may be caused by the reason of increased body weight, alcohol consumption, gastroesophageal reflux disease and premalignant. In western countries, the 5-year rate of advanced AEG was less than 30%, it was the same in China. There was significant difference in epidemiology, pathogenic mechanism, biological characteristics and prognosis between AEG and antrum tumors, so AEG was regarded as a kind of independent disease. Up till now, the scope of lymph node dissected, the selection of operation approach, the resection range and the digestive tract reconstruction for the treatment of AEG were in dispute, especially in the reconstruction of digestive tract after operation. The purpose of this study is to investigate the efficacy and safety of the proximal gastrectomy combined with Giraffe anastomosis for early adenocarcinoma of esophagogastric junction.

DETAILED DESCRIPTION:
In the past years, the adenocarcinoma of the esophagogastric junction (AEG) has been increasing obviously in China. It may be caused by the reason of increased body weight, alcohol consumption, gastroesophageal reflux disease and premalignant. In western countries, the 5-year rate of advanced AEG was less than 30%, it was the same in China. There was significant difference in epidemiology, pathogenic mechanism, biological characteristics and prognosis between AEG and antrum tumors, so AEG was regarded as a kind of independent disease. Up till now, the scope of lymph node dissected, the selection of operation approach, the resection range and the digestive tract reconstruction for the treatment of AEG were in dispute, especially in the reconstruction of digestive tract after operation.

The digestive tract reconstruction methods for AEG II were determined by the surgical approach. The controversy exists regarding whether reconstruction method with low esophageal reflux should be used to treat AEG patients. The gastric tube reconstruction, the antrum-preserving double-tract reconstruction and the Roux-en-Y reconstruction were the common methods. Some studies showed that the 24-h pH profile in the patients with gastric tube reconstruction was similar to the healthy person, but it may be related to the increasing incidence of gastroesophageal reflux disease in the healthy person and the anti-reflux medication used in the patients. Although the antrum-preserving double-tract reconstruction have a good function of anti-reflux, the complicated operation and too many anastomotic stomas increased the rate of postoperative happened. The common physiological mechanism of anti-reflux was caused by the lower esophageal sphincter, esophagogastric junction, His angle and so on. Therefore, in our center, we use a new reconstruction which combine the advantages of gastric tube reconstruction with rebuilding the His angle and fundus of gastric. We call it Gastric tube interposition esophagogastrostomy with reconstruction of His angle and fundus (Giraffe anastomosis).

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative endoscopy and biopsy confirmed adenocarcinoma of esophagogastric junction, and predictively feasible of transabdominal proximal gastrectomy.
2. Early gastric cancer, of preoperative staging AJCC 8th Edition cT1N0M0 and not suitable for endoscopic resection;
3. Completion of abdominal CT scan and ultrasound endoscopy
4. Age：18 to 70 years ;
5. Karnofsky score ≥ 70
6. With good compliance and informed consent required.

Exclusion Criteria:

1. Pregnancy, breast-feeding women.
2. The existence of the peripheral nervous system disorders or significant neurological disorders and a history of central nervous system disorders.
3. Severity mental diseases;
4. Patients with other severe complications cannot tolerate surgery: such as severe heart and lung diseases, heart function below clinical stage 2, uncontrollable hypertension, pulmonary infection, moderate to severe COPD, chronic bronchitis, severe diabetes and / or renal insufficiency, severe hepatitis and / or function below the rank of CHILD B grade, and severe malnutrition, etc.
5. With other malignancies which were not cured.
6. Patients have already joined other clinical trials
7. After signature the Clinical trial agreement, patients and their agent will quit the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Rate of reflux esophagitis after operation | 12 months
  The rate of reflux esophagitis after operation will be assessed by gastrointestinal endoscopy with Los Angeles (LA) classification and the reflux disease questionnaire (RDQ) scores were used to evaluate postoperative gastroesophageal reflux.

SECONDARY OUTCOMES:
Postoperative quality of life: European Organization for Research and Treatment of Cancer (EORTC) | 12 months
  Assessed by European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) - C30 questionnaire, the total score ranges from 30 to 126, and higher values represent a worse outcome.
Postoperative recovery | 12 months
  postoperative complication rate according to the Clavian-Dindo classification, postoperative death rate with 30 days
Postoperative nutrition status | 12months
  Change of Hemoglobin, Vitamin B12 cumulative supplement quantity

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital), Hangzhou, Zhejiang, China